CLINICAL TRIAL: NCT06660225
Title: Towards Closed Loop Deep Brain Stimulation for Treatment of Refractory Obsessive-Compulsive Disorder
Brief Title: Deep Brain Stimulation for Refractory Obsessive-Compulsive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nader Pouratian (Other)
Responsible Party: Sponsor-Investigator, Nader Pouratian, Professor and Chair, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2024-0733
Record Dates: First submitted 2024-10-05; First posted 2024-10-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive; Compulsive; Deep Brain Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: There will be two 4 month blocks in which, depending on group assignment, participants will receive either active or sham stimulation from the DBS device. Following completing of the first 4 month block, the groups will cross-over. Individuals originally receiving active stimulation will now receive sham, and individuals receiving sham stimulation originally will now receive active stimulation. Following the completing of both four month blocks, all participants will receive active open-label treatment. Continued follow-up psychiatric assessments will be preformed every two week during the double-blind portion of the trial, and then every 6 weeks during the open-label treatment phase.
Who Masked: Participant, Investigator
Masking Description: Neither the participant of investigator will know which treatment group an individual is assigned to. After the completion of the blinded portion of the trial, all participants will be transitioned to open-label stimulation/treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Sham Control stimulation, then Therapeutic stimulation (Experimental): Subject randomized to this arm are initially "OFF" DBS (Deep Brain Stimulation) prior to the open label period for 16 weeks and then "ON" DBS for the next 16 weeks. This is then followed by an open-label period of DBS stimulation.
  Interventions: Device: Medtronic Percept Deep Brain Stimulation Therapy [Sham Control Stimulation]; Device: Medtronic Percept Deep Brain Stimulation Therapy [Therapeutic stimulation]
- Therapeutic stimulation, then Sham Control stimulation (Experimental): Subjects randomized to this arm are initially "ON" DBS prior to the open label period for 16 weeks and then "OFF" DBS for the next 16 weeks. This is followed by an open-label stimulation period.
  Interventions: Device: Medtronic Percept Deep Brain Stimulation Therapy [Sham Control Stimulation]; Device: Medtronic Percept Deep Brain Stimulation Therapy [Therapeutic stimulation]
- Therapeutic stimulation (Experimental): All participants will transition to an open label stimulation phase for chronic therapy after the cross-over portion of this trial
  Interventions: Device: Medtronic Percept Deep Brain Stimulation Therapy [Therapeutic stimulation]

INTERVENTIONS:
Device: Medtronic Percept Deep Brain Stimulation Therapy [Sham Control Stimulation] — Deep brain stimulation is a surgery where bilateral electrodes are precisely inserted to specific brain targets affected by a disease state, and electrical stimulation is applied to achieve symptom relief. DBS is a reversible and adjustable treatment option and is now a preferred alternative to neurosurgical ablation. Sham Stimulation=DBS OFF
  Arms: Sham Control stimulation, then Therapeutic stimulation; Therapeutic stimulation, then Sham Control stimulation
Device: Medtronic Percept Deep Brain Stimulation Therapy [Therapeutic stimulation] — Deep brain stimulation is a surgery where bilateral electrodes are precisely inserted to specific brain targets affected by a disease state, and electrical stimulation is applied to achieve symptom relief. DBS is a reversible and adjustable treatment option and is now a preferred alternative to neurosurgical ablation. Therapeutic Stimulation= DBS ON

SUMMARY:
The goal of this clinical trial is to learn if deep brain stimulation (DBS) works to treat refractory obsessive-compulsive disorder (OCD). The main questions it aims to answer are:

* Assess the effects of the anteromedial sub-thalamic nucleus (amSTN)stimulation on obsessive/compulsive symptoms.
* Map the amSTN using neuronal responses [single unit and local field potentials (LFP) recordings] at rest and under high frequency stimulation during surgery.
* Record chronic brain activity with the implanted pulse generator and look for neuronal signatures correlated with symptom severity.

Researchers will compare active deep brain stimulation to a placebo (sham stimulation) to see if DBS works to treat refractory OCD.

Participants will:

* Undergo surgery for the implantation of a deep brain stimulation device
* Follow-up visits every three weeks with study staff
* 6 month follow-up for the next 2-3 years after first year of study participation is complete

DETAILED DESCRIPTION:
The primary goal of this research study is to conduct a small scale randomized, double-blind clinical cross-over trial of deep brain stimulation for obsessive-compulsive disorder targeting the anteromedial subthalamic nucleus (amSTN), with which study team will not only produce high quality data of the clinical efficacy of DBS for OCD, but also attain critical insights into the neurophysiological underpinnings of disease and symptoms in OCD. This work will support future innovative therapy development, including refinement of surgical targeting and optimization of therapeutic stimulation.

This will be a 3-year study with the aim of implanting 10 patients with bilateral amSTN DBS leads. Intra-operatively, precise single neuron recordings will be obtained at the therapeutic target while the patient participates symptom provocation. Participants will be implanted with a sensing pulse generator (Medtronic Percept) which enables chronic recordings from the amSTN target in addition to providing therapeutic stimulation. Each participant will be randomized to start with either a sham control stimulation phase or therapeutic stimulation, and cross-over at 4 months. If symptoms recur upon cross-over from therapeutic to sham stimulation, participants will exit the sham stimulation phase and rescue therapy/stimulation will be delivered. All participants will transition to an open label stimulation phase for chronic therapy. Multiple assessments of the participants will follow, including OCD severity, cognition, behavior, and side effects.

Formal psychiatric assessments will take place at two weeks, at one month, and then once every three weeks during the randomization blinded period and then every 6 weeks during the open label period. During psychiatric assessments, the PERCEPT device will be used to obtain neural recordings of the STN activity.

Additionally, for the secondary outcome measure for the association between amSTN activity and cognitive/emotional measure there are two components of this measure that are of a qualitative nature. Burstiness and coherence are unitless measures and thus will not be included in the outcome measure reporting section. They will instead be discussed in the limitation section at annual reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of obsessive-compulsive disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria
* Severe OCD assessed by the Yale-Brown Obsessive-Compulsive Scale (YBOCS) with a score of more than 27
* Refractory OCD; severe symptoms and impairment for more than 5 years despite pharmacological and psychological treatment.
* Have failed to improve following treatment with at least two serotonin transport inhibitors and one augmenting agent taken for an adequate time period.
* Having failed to improve despite adequate cognitive behavioral therapy, as evaluated by the study psychiatrist
* Patients between 22 and 75.
* Ability to understand and sign written informed consent by the patient.

Exclusion Criteria:

* Diagnosis of severe major depression disorder (MDD) with psychotic features.
* Significant suicidal risk [Hamilton Depression scale item 3 (suicide)>2].
* Comorbidity with any primary Psychotic Disorder, Post-Traumatic Stress Disorder (PTSD), or Eating Disorder.
* History of substance or alcohol dependence or abuse in the preceding 12 months.
* Significant cognitive decline, measured by Mini-Mental State Examination (MMSE <26) and Montreal Cognitive Assessment (MoCA; <24).
* Any other current clinical significant neurological disorder or medical illness affecting brain function, other than a tic disorder.
* Any clinically significant abnormality on preoperative MRI that would affect the safety of the surgical procedure in the opinion of the study neurosurgeon.
* Any DBS contraindication, infection, coagulopathy, significant cardiac risk factors, or other medical risk factors for surgery.
* Pregnancy.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of amSTN stimulation on OCD symptoms as measured by YBOCS | 36 months
  Assessment of the efficacy of amSTN stimulation on OCD symptoms. This will be assessed by the Yale-Brown Obsessive-Compulsive Scale (YBOCS). Possible scores range from 0-5 where lower scores indicate better outcome.
Incidence of Adverse events | 36 months
  Safety will be assessed with cumulative serious adverse event rate that will be Frequency at which AEs occur that are directly related to the study device.

SECONDARY OUTCOMES:
Effect of DBS on Mood and Quality of Life as measured by HAM-A survey | 36 months
  Hamilton Scale for Anxiety. A rating scale developed to measure the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and semantic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score ranger of 0-56, where 17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Effect of DBS on Mood and Quality of Life as measured by HAM-D21 survey | 36 months
  Hamilton Depression Rating Scale (HAM-D). A 21-item version of the HAM-D that includes 4 items intended to subtype the depression. The HAM-D is originally a 17 item questionnaire pertaining to symptoms of depression experienced over the past week. The patients score is determined using the first 17 questions. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial. Scoring on each question varies.
Effect of DBS on Mood and Quality of Life as measured by BPRS survey | 36 months
  Brief Psychiatric Rating Scale (BPRS). An assessment that assesses the level of the following symptoms; somatic concern, anxiety, emotional withdrawal, conceptual disorganization, guilt feelings, tension, mannerisms and posturing, grandiosity, depressive mood, hostility, suspiciousness, hallucinatory behavior, motor retardation, uncooperativeness, unusual thought content, blunted affect, excitement, disorientation. Items are scored on a 1(not present) to 7 (extremely severe) scale. It is based on the clinicians interview with the patients and observations of the patient behavior over the previous 2-3 days.
Effect of DBS on Mood and Quality of Life as measured by CGI-S survey | 36 months
  Clinical Global Inventory- Severity scale is used to measure this outcome (CGI-S). This is a 3-item observer-rated scale that measures illness severity (CGI-S). The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through 7 (amongst the most severely ill patients).
Effect of DBS on Mood and Quality of Life as measured by MMSE tool | 36 months
  Mini-Mental State Examination (MMSE). A questionnaire comprised of 11 questions that is used by doctors and other health professionals to check for cognitive impairment. It is typically used to see if you have problems with ones thinking or communication. It can check for problems with understanding and amnesia. The MMSE checks 6 areas of mental ability including; knowing when one is (date and place), attention and concentration, short-term memory (recall), language skills, visual and spatial relationship between objects, ability to understand and follow instructions. The assessment is scored out of 30. A score of 25 or higher is normal, and score below 24 could indicate cognitive impairment.
Association between amSTN activity and cognitive/emotional measures as measured by rate of neural activity | 36 months
  The rate of neural activity will be measured via Hz.
Association between amSTN activity and cognitive/emotional measures as measured by amplitude of neural activity | 36 months
  Amplitude of neural activity will be measured via microamps.
Association between amSTN activity and cognitive/emotional measures as measured by phase | 36 months
  A unit of measurement used to quantify the relationship between the temporal structures of signals in the brain, and are often used to study functional connectivity in neuroscience. This outcome measure will be measured in units of 0-2π.
Association between amSTN activity and cognitive/emotional measures as measured by cross-frequency coupling of neural activity. | 36 months
  Cross-frequency coupling (CFC) is a neuroscience measure that describes the statistical relationship between the frequency, amplitude, or phase of two different frequency bands in the brain. Its a type of neural oscillatory coupling that is been studied in the context of brain health and disease. This data point will be measured via the modulation index.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Pouratian, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Investigators with established research programs will be eligible for data sharing. Interested investigators will be required to submit a summary of proposed work and requested data elements. If approved by the Principal Investigator of the study, data will be shared. This data will be de-identified and coded. There is no plan to share identifiers outside the study team.